CLINICAL TRIAL: NCT02855437
Title: Novel Methods for Ascertainment of Gout Flares -A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Vice Chair, Department of Medicine; Jane Knight Lowe Professor, Division of Clinical Immunology and Rheumatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: X160105005; ESR-15-11070 (Other: AstraZenca)
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Voice Response (Active Comparator): The interactive voice response system (IVR) is an automated telephone system that is used to contact study participants. At enrollment the study coordinator will explain how the IVR works, planned survey schedule, and that participant -initiated calls to IVR are allowed.
  Interventions: Device: IVR (Phone call)
- RheumPro Smartphone Application (Active Comparator): RheumPro is a UAB developed smartphone application to capture patient reported outcomes. At enrollment the study coordinator will explain how RheumPro works, planned survey schedule, and that participant -initiated surveys in RheumPro are allowed.
  Interventions: Device: RheumPro (Smartphone application)

INTERVENTIONS:
Device: IVR (Phone call) — IVR will auto dial participants at a schedule time. Participants complete questions using their phone keypad. Participants can also call the IVR to complete surveys if they experience a flare. The IVR will be programmed to call the patient weekly for 26 weeks to complete a weekly Gout Flare Survey and Patient Reported Outcomes Survey. Consistent with the published gout flare self-report definition, gout flare ascertainment questions will include whether the recent flare is similar to past flares, the number of swollen joints and the number of warm joints. Pain at rest during the attack will be assessed on a 0-9 scale. Further questions will include peak pain, timing of attack and duration of attack if completed. We will capture patient reported outcome measures (e.g. pain, fatigue, sleep) using instruments from NIH PROMIS. Following completion of 26 week IVR period participants will crossover to RheumPro arm.
  Arms: Interactive Voice Response
Device: RheumPro (Smartphone application) — RheumPRO will be programmed to notify participants weekly for 26 weeks via a scheduled "pop-up" to complete Gout Flare and Patient Reported Outcomes Surveys. Participants self-navigate through the survey questions using their smartphone. If participants do not complete the Gout Flare or Patient Reported Outcomes surveys RheumPro will generate 2 more "pop-ups" at the same time over the proceeding 2 days (eg. Tuesday 4 PM, Wednesday 4 PM). Participants can also open the RheumPro application on their smartphone and complete surveys or if they experience a flare on a day they are not scheduled to complete a survey. Following completion of 26 week RheumPro period participants will crossover to IVR arm.
  Arms: RheumPro Smartphone Application

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of using different remote data collection technologies to ascertain flare occurrence among gout patients. Two technologies will be the focus of this study: a telephone based interactive voice response (IVR) and a smartphone mobile application (called RheumPRO). The results of this study will not only guide research approaches in clinical trials, but may also have direct implications for monitoring patient outcomes in the context of day-to-day clinical practice.

The investigators hypothesize that acceptability will be greater for RheumPRO application than IVR. Additionally, the investigators hypothesize that RheumPRO will be associated with a greater frequency of patient-initiated interactions.

DETAILED DESCRIPTION:
Acute gout flares are a major cause of morbidity. Flares lead to substantial reductions in health-related quality of life, increased work absenteeism, productivity loss, and substantial healthcare costs. Acute gout flares are likely related to more than 174,000 emergency department visits in the U.S. annually with corresponding charges approaching $166 million.

In recent surveys, gout patients and healthcare providers alike identified the reduction of gout flares as the highest priority outcome that should be examined in future comparative effectiveness studies of urate lowering therapy (ULT) (unpublished results). Despite consensus about the importance of capturing flares, clinical trials investigating ULTs or anti-inflammatory prophylaxis have used inconsistent flare definitions and methods of flare ascertainment. The inconsistency has likely been driven by the absence of a standardized definition or ascertainment method. These deficits limit comparisons that can be made across investigations.

Recently, a group supported by the American College of Rheumatology & European League Against Rheumatism (ACR & EULAR) has attempted to define a gout flare (8-10). For simplicity, the group focused on defining only those flares occurring after a definitive gout diagnosis. Nine elements of a flare definition emerged from the first two studies. These nine elements included physician reported information, laboratory data and patient self-report. In a third study, Gaffo et al. compared the discriminatory ability of the self-reported items against the gold standard of a rheumatologist's judgment of flare presence. Self-report of 4 criteria had the greatest discriminatory ability with an area under the curve (AUC) of 0.931. These promising results indicate the important role for a standardized self-report definition of a gout flare.

In addition to variability in gout flare definitions, the optimal method for obtaining self-reported flares remains undefined. An early study of febuxostat, for example, assessed flares weekly at physician visits Another study counted a flare only when it was treated by a healthcare provider. Still other studies assessed flares during physician visits occurring at variable time points. These inconsistent methods also pose practical limitations given by their time and resource intensive nature. Opportunities to increase efficiency have only recently become available with the validation of the self-reported definition for gout flares described above. Self-report can now be combined with technological advances in remote data collection to develop novel and highly efficient methods to identify gout flares. The investigators propose a study to address this pressing need by leveraging technological advances that facilitate the remote and real-time collection of patient reported flares and outcomes (PROs) in gout.

ELIGIBILITY:
Inclusion Criteria:

* >/= to 18 yrs of age with Current physician diagnosed gout
* current hyperuricemia (serum urate level >6.8 mg/dl)
* self-report of at least two gout flares in the previous 6 months
* current smartphone user utilizing a FitBit compatible smart Phone (with the ability to download RheumPRO from Apple/Google Play store).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Saag, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg R, Sayles HR, Yu F, Michaud K, Singh J, Saag KG, Mikuls TR. Gout-related health care utilization in US emergency departments, 2006 through 2008. Arthritis Care Res (Hoboken). 2013 Apr;65(4):571-7. doi: 10.1002/acr.21837. PMID 22949176
- [Background] Becker MA, Schumacher HR Jr, Wortmann RL, MacDonald PA, Palo WA, Eustace D, Vernillet L, Joseph-Ridge N. Febuxostat, a novel nonpurine selective inhibitor of xanthine oxidase: a twenty-eight-day, multicenter, phase II, randomized, double-blind, placebo-controlled, dose-response clinical trial examining safety and efficacy in patients with gout. Arthritis Rheum. 2005 Mar;52(3):916-23. doi: 10.1002/art.20935. PMID 15751090
- [Background] Becker MA, Schumacher HR Jr, Wortmann RL, MacDonald PA, Eustace D, Palo WA, Streit J, Joseph-Ridge N. Febuxostat compared with allopurinol in patients with hyperuricemia and gout. N Engl J Med. 2005 Dec 8;353(23):2450-61. doi: 10.1056/NEJMoa050373. PMID 16339094
- [Background] Schumacher HR Jr, Becker MA, Wortmann RL, Macdonald PA, Hunt B, Streit J, Lademacher C, Joseph-Ridge N. Effects of febuxostat versus allopurinol and placebo in reducing serum urate in subjects with hyperuricemia and gout: a 28-week, phase III, randomized, double-blind, parallel-group trial. Arthritis Rheum. 2008 Nov 15;59(11):1540-8. doi: 10.1002/art.24209. PMID 18975369
- [Background] Becker MA, Schumacher HR, Espinoza LR, Wells AF, MacDonald P, Lloyd E, Lademacher C. The urate-lowering efficacy and safety of febuxostat in the treatment of the hyperuricemia of gout: the CONFIRMS trial. Arthritis Res Ther. 2010;12(2):R63. doi: 10.1186/ar2978. Epub 2010 Apr 6. PMID 20370912
- [Background] Sundy JS, Baraf HS, Yood RA, Edwards NL, Gutierrez-Urena SR, Treadwell EL, Vazquez-Mellado J, White WB, Lipsky PE, Horowitz Z, Huang W, Maroli AN, Waltrip RW 2nd, Hamburger SA, Becker MA. Efficacy and tolerability of pegloticase for the treatment of chronic gout in patients refractory to conventional treatment: two randomized controlled trials. JAMA. 2011 Aug 17;306(7):711-20. doi: 10.1001/jama.2011.1169. PMID 21846852
- [Background] Borstad GC, Bryant LR, Abel MP, Scroggie DA, Harris MD, Alloway JA. Colchicine for prophylaxis of acute flares when initiating allopurinol for chronic gouty arthritis. J Rheumatol. 2004 Dec;31(12):2429-32. PMID 15570646
- [Background] Taylor WJ, Schumacher HR Jr, Baraf HS, Chapman P, Stamp L, Doherty M, McQueen F, Dalbeth N, Schlesinger N, Furst DE, Vazquez-Mellado J, Becker MA, Kavanaugh A, Louthrenoo W, Bardin T, Khanna D, Simon LS, Yamanaka H, Choi HK, Zeng X, Strand V, Grainger R, Clegg D, Singh JA, Diaz-Torne C, Boers M, Gow P, Barskova VG. A modified Delphi exercise to determine the extent of consensus with OMERACT outcome domains for studies of acute and chronic gout. Ann Rheum Dis. 2008 Jun;67(6):888-91. doi: 10.1136/ard.2007.079970. Epub 2007 Nov 29. PMID 18055475
- [Background] Taylor WJ, Shewchuk R, Saag KG, Schumacher HR Jr, Singh JA, Grainger R, Edwards NL, Bardin T, Waltrip RW, Simon LS, Burgos-Vargas R. Toward a valid definition of gout flare: results of consensus exercises using Delphi methodology and cognitive mapping. Arthritis Rheum. 2009 Apr 15;61(4):535-43. doi: 10.1002/art.24166. PMID 19333981
- [Background] Gaffo AL, Schumacher HR, Saag KG, Taylor WJ, Dinnella J, Outman R, Chen L, Dalbeth N, Sivera F, Vazquez-Mellado J, Chou CT, Zeng X, Perez-Ruiz F, Kowalski SC, Goldenstein-Schainberg C, Chen L, Bardin T, Singh JA. Developing a provisional definition of flare in patients with established gout. Arthritis Rheum. 2012 May;64(5):1508-17. doi: 10.1002/art.33483. PMID 22083456
- [Derived] Elmagboul N, Coburn BW, Foster J, Mudano A, Melnick J, Bergman D, Yang S, Chen L, Filby C, Mikuls TR, Curtis JR, Saag K. Physical activity measured using wearable activity tracking devices associated with gout flares. Arthritis Res Ther. 2020 Aug 3;22(1):181. doi: 10.1186/s13075-020-02272-2. PMID 32746893
- [Derived] Elmagboul N, Coburn BW, Foster J, Mudano A, Melnick J, Bergman D, Yang S, Redden D, Chen L, Filby C, Curtis JR, Mikuls TR, Saag KG. Comparison of an interactive voice response system and smartphone application in the identification of gout flares. Arthritis Res Ther. 2019 Jun 29;21(1):160. doi: 10.1186/s13075-019-1944-5. PMID 31255174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population recruited was patients with gout. Patients were recruited from the UAB gout clinic, The Kirklin Clinic, and the UNMC gout clinic.
Groups:
- Interactive Voice Response, Then RheumPRO: IVR will auto dial participants at a schedule time. Participants complete questions using their phone keypad. Participants can also call the IVR to complete surveys if they experience a flare. The IVR will be programmed to call the patient weekly for 26 weeks to complete a weekly Gout Flare Survey and Patient Reported Outcomes Survey. Consistent with the published gout flare self-report definition, gout flare ascertainment questions will include whether the recent flare is similar to past flares, the number of swollen joints and the number of warm joints. Pain at rest during the attack will be assessed on a 0-9 scale. Further questions will include peak pain, timing of attack and duration of attack if completed. We will capture patient reported outcome measures (e.g. pain, fatigue, sleep) using instruments from NIH PROMIS. Following completion of 26 week IVR period participants will crossover to RheumPro arm.
- RheumPro Smartphone Application, Then IVR: RheumPRO will be programmed to notify participants weekly for 26 weeks via a scheduled "pop-up" to complete Gout Flare and Patient Reported Outcomes Surveys. Participants self-navigate through the survey questions using their smartphone. If participants do not complete the Gout Flare or Patient Reported Outcomes surveys RheumPro will generate 2 more "pop-ups" at the same time over the proceeding 2 days (eg. Tuesday 4 PM, Wednesday 4 PM). Participants can also open the RheumPro application on their smartphone and complete surveys or if they experience a flare on a day they are not scheduled to complete a survey. Following completion of 26 week RheumPro period participants will crossover to IVR arm.
Period: Phase 1
Arm/Group | Interactive Voice Response, Then RheumPRO | RheumPro Smartphone Application, Then IVR
Started | 23 | 21
Completed | 21 | 19
Not Completed | 2 | 2
Period: Crossover Period (Same Day)
Arm/Group | Interactive Voice Response, Then RheumPRO | RheumPro Smartphone Application, Then IVR
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | Interactive Voice Response, Then RheumPRO | RheumPro Smartphone Application, Then IVR
Started | 21 | 19
Completed | 20 | 18
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of participants completing the study (N = 44)
Groups:
- Overall: Overall description of participants in the pilot study entitled, "Novel Methods for Ascertainment of Gout Flares -A Pilot Study"
Arm/Group | Overall
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White race | 30
  Race: Black or other race | 14
Age of first gout flare [Mean (Standard Deviation); unit: Years] | 38.3 (18.6)
Number of flares prior 6 months [Count of Participants; unit: Participants]
  2-3 flares in prior 6 months | 19
  >=4 flares in prior 6 months | 25

OUTCOME MEASURES:

1. Primary Outcome: Preference IVR vs RheumPRO
Description: Percentage of total study population preferring IVR vs. RheumPRO
Time Frame: 6 months
Population: Preference of IVR and StudyBuddy for reporting gout flares as reported by participants
Measure: Count of Participants; unit: Participants
Groups:
- Interactive Voice Response: The interactive voice response system (IVR) is an automated telephone system that is used to contact participants. At enrollment the study coordinator will explain how the IVR works, planned survey schedule, and that participant -initiated calls to IVR are allowed.
  IVR (Phone call): IVR will auto dial participants at a schedule time. Participants complete questions using their phone keypad. Participants can also call the IVR to complete surveys if they experience a flare. The IVR will be programmed to call the patient weekly for 26 weeks to complete a weekly Gout Flare Survey and Patient Reported Outcomes Survey. Consistent with the published gout flare self-report definition, gout flare ascertainment questions will include whether the recent flare is similar to past flares, the number of swollen joints and the number of warm joints. Pain at rest during the attack will be assessed on a 0-9 scale. Further questions will include peak pain, timing of attack and duration of attack
- RheumPro Smartphone Application: RheumPro is a UAB developed smartphone application to capture patient reported outcomes. At enrollment the study coordinator will explain how RheumPro works, planned survey schedule, and that participant -initiated surveys in RheumPro are allowed.
  RheumPro (Smartphone application): RheumPRO will be programmed to notify participants weekly for 26 weeks via a scheduled "pop-up" to complete Gout Flare and Patient Reported Outcomes Surveys. Participants self-navigate through the survey questions using their smartphone. If participants do not complete the Gout Flare or Patient Reported Outcomes surveys RheumPro will generate 2 more "pop-ups" at the same time over the proceeding 2 days (eg. Tuesday 4 PM, Wednesday 4 PM). Participants can also open the RheumPro application on their smartphone and complete surveys or if they experience a flare on a day they are not scheduled to complete a survey. In addition RheumPro questionnaires at months 1 , 3, and 6 will assess RheumPro ease of use.
Arm/Group | Interactive Voice Response | RheumPro Smartphone Application
Number analyzed (Participants) | 38 | 38
Participants | 3 | 28

2. Primary Outcome: Feasibility of Using IVR vs. RheumPRO to Report Gout Flares
Description: Feasibility ----Assessed by the percentage of participants completing answer IRV/RheumPRO queries.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of weekly response
Groups:
- RheumPro Smartphone Application: RheumPro is a UAB developed smartphone application to capture patient reported outcomes. At enrollment the study coordinator will explain how RheumPro works, planned survey schedule, and that participant -initiated surveys in RheumPro are allowed.
  RheumPro (Smartphone application): RheumPRO will be programmed to notify participants weekly for 26 weeks via a scheduled "pop-up" to complete Gout Flare and Patient Reported Outcomes Surveys. Participants self-navigate through the survey questions using their smartphone. If participants do not complete the Gout Flare or Patient Reported Outcomes surveys RheumPro will generate 2 more "pop-ups" at the same time over the proceeding 2 days (eg. Tuesday 4 PM, Wednesday 4 PM). Participants can also open the RheumPro application on their smartphone and complete surveys or if they experience a flare on a day they are not scheduled to complete a survey. In addition RheumPro questionnaires at months 1 , 3, and 6 will assess RheumPro ease of use,
Arm/Group | Interactive Voice Response | RheumPro Smartphone Application
Number analyzed (Participants) | 38 | 38
percentage of weekly response | 81 (21) | 80 (25)

ADVERSE EVENTS:
Time Frame: AE data were not collected in this study.
Description: AE data were not collected in this study.
Arm/Group | Interactive Voice Response | RheumPro Smartphone Application
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02855437/Prot_SAP_000.pdf